CLINICAL TRIAL: NCT04566445
Title: HORIZON: A Phase II, Open-label, Outcomes-assessor Masked, Multicentre, Randomised, Controlled Study to Evaluate the Safety and Efficacy of Two Doses of GT005 Administered as a Single Subretinal Injection in Subjects With Geographic Atrophy Secondary to Dry Age-related Macular Degeneration
Brief Title: HORIZON: A Phase II Study to Evaluate the Safety and Efficacy of Two Doses of GT005
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for interim analysis demonstrating futility (trial highly unlikely to meet efficacy outcome). The trial is not ending early because of medical problems or concerns.
Sponsor: Gyroscope Therapeutics Limited (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT005-03; CPPY988A12201 (Other: Novartis); 2020-002431-30 (EudraCT Number)
Record Dates: First submitted 2020-09-09; First posted 2020-09-28 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: Dry age-related macular degeneration; Geographic atrophy; Retinal disease; Eye disease; Retinal degeneration; Macular atrophy
MeSH Terms: conditions — Geographic Atrophy; Retinal Diseases; Eye Diseases; Retinal Degeneration; Anetoderma

STUDY DESIGN:
Intervention Model Description: This is a Phase II, open-label, outcomes-assessor masked, multicentre, randomised, controlled study to evaluate the safety and efficacy of two doses of GT005 administered as a single subretinal injection in subjects with GA secondary to AMD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcome Assessor). The overall objectives of the study are to evaluate the safety and efficacy (anatomical and functional visual outcomes) of two doses of GT005 in genetically defined subjects with GA due to AMD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GT005 Medium dose [5E10 vg] (Experimental): GT005 Medium dose [5E10 vg]
  Interventions: Drug: GT005
- GT005 High dose [2E11 vg] (Experimental): GT005 High dose [2E11 vg]
  Interventions: Drug: GT005
- Untreated control (No Intervention): Untreated control

INTERVENTIONS:
Drug: GT005 — GT005 is a recombinant, non-replicating AAV2 expressing human complement factor I (CFI). GT005 was administered as a single time subretinal injection into the study eye of subjects allocated to one of the two GT005 doses.
  Arms: GT005 High dose [2E11 vg]; GT005 Medium dose [5E10 vg]

SUMMARY:
The purpose of this clinical study was to evaluate the safety and efficacy of two doses of GT005 administered as a single subretinal injection in subjects with geographic atrophy secondary to age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This was a Phase II, open-label, outcomes-assessor masked, multicenter, randomized, controlled study designed to evaluate the safety and efficacy of two doses of GT005 administered as a single-time subretinal injection in subjects with Geographic atrophy (GA) secondary to Age-related macular degeneration (AMD).

Approximately 250 subjects, across Stage 1 and Stage 2, were planned to be randomized to one of two doses of GT005 or the untreated control group.

Subjects entered the study had genotyping and serum Complement factor I (CFI) levels assessed either through participation in a previous Gyroscope sponsored study, or a Sponsor-approved laboratory during the HORIZON screening period. If both eyes are eligible; the eye with the worse visual acuity will be selected as the study eye. If subjects failed to meet the eligibility criteria for this study, they were classified as screen failures and could be considered for entry into another Novartis/Gyroscope sponsored study.

After providing the informed consent, subjects underwent ophthalmic and clinical assessments to determined eligibility for inclusion in the study.

Upon confirmation of eligibility, subjects were randomized to one of two dose groups (medium dose [5E10 vg] or high dose [2E11 vg]). Within each dose group, subjects were allocated to GT005, or untreated control based on a 2:1 ratio. The overall study population (N=approximately 250) aimed to include approximately 60% of subjects with foveal GA and 40% of subjects with non-foveal GA (extrafoveal lesions). The study eye was identified for all subjects.

Enrolment for HORIZON were composed of two stages. Stage 1 enrolled subjects with foveal or non-foveal GA until 180 subjects were randomized. Stage 2 enrolled subjects with nonfoveal GA. Subjects with a CFI rare variant associated with normal or low serum CFI were also allowed to be enrolled in Stage 2, irrespective of GA foveal involvement.

Subjects were stratified by GA lesion size on Fundus autofluorescence (FAF) (≤10 mm2 or >10 mm2) and AMD genotype subgroup. Randomization of study eyes in the GA lesion size upper stratum of >10 mm2 to 17.5 mm2 was capped at 20% of total subjects randomized in Stage 1 and Stage 2, respectively. In Stage 2, once enrolment capping at 20% based on upper GA lesion size was reached, eyes that fulfilled the cap criteria were no longer eligible, unless the subject had a CFI rare variant genotype (minor allele frequency ≤1%) previously associated with normal or low serum CFI or had an unreported CFI rare variant genotype (Group 1 and 5). A permuted-block method was used to obtain an approximately 2:1 ratio between GT005 and the untreated control groups for each dose group within each stratum.

Following randomization, the Investigator was informed of the subject's allocated treatment (GT005 or the untreated control group) and the study eye selected. To minimize bias during imaging grading, all imaging endpoint assessments and grading were performed at a Central reading centre (CRC). All imaging efficacy assessments were performed in a masked fashion. The Sponsor, subjects, investigators, and study personnel performing clinical assessments remained masked to the dose received for those allocated to GT005.

For each subject, the study comprised of a screening period lasting up to 8 weeks (or up to 12 weeks if agreed by the Sponsor Medical Monitor) followed by a 96-week study period. All subjects were assessed for the occurrence of AEs at each visit and underwent functional assessments, retinal imaging, and biological sampling as per the schedule of assessments.

This study was conducted in compliance with Independent ethics committees (IECs) / Institutional review boards (IRBs), informed consent regulations, the Declaration of Helsinki, International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP) Guidelines, and the Food and Drug Administration (FDA), 21 Code of Federal Regulations (CFR) Part 11, Electronic Records, Electronic Signatures, and FDA, Guidance for Industry: Computerised Systems Used in Clinical Trials.

On 24-Aug-2023, the decision was taken to terminate the study and the GT005 program. The decision was aligned with the recommendation of an independent Data monitoring committee (DMC), which concluded that futility criteria had been met for the HORIZON study (GT005-03) and the overall benefit-risk ratio did not support continuation of the current development program as planned. All GT005- treated subjects, who were willing to be transferred into the long-term safety follow-up study were enrolled in the ORACLE (CPPY988A12203B) study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent
2. Age ≥55 years
3. a. In Stage 1: Have a clinical diagnosis of GA secondary to AMD in the study eye, as determined by the Investigator, and a diagnosis of AMD in the contralateral eye; b. In Stage 2: Have a clinical diagnosis of GA secondary to AMD in the study eye, as determined by the Investigator, that is non-foveal, as determined by the central reading centre, or has a CFI rare variant genotype and meets inclusion criteria 3a, and a diagnosis of AMD in the contralateral eye (except if monocular)
4. GA lesion(s) within an acceptable size on FAF, in the study eye
5. The GA lesion in the study eye must reside completely within the FAF image
6. Up to 25% of the enrolled study population are permitted to have CNV in the fellow eye
7. Have a BCVA of ≥24 letters (6/95 or 20/320 Snellen acuity equivalent), using ETDRS charts, in the study eye
8. a. In Stage 1: Meet one of the pre-specified AMD genetic subgroup criteria; b. In Stage 2: Genotyping is not required for study eligibility
9. Able to attend all study visits and complete the study procedures
10. Women of child-bearing potential must have a negative pregnancy test within 2 weeks prior to randomisation (not required for postmenopausal women) or provide documentation of being surgically sterilised

Exclusion Criteria:

1. a. In Stage 1: Carriers of excluded genetic variants; b. In Stage 2: Subjects are excluded if they have a clinical diagnosis of Stargardt Disease or other retinal dystrophies
2. Have a history, or evidence, of CNV in the study eye
3. Presence of moderate/severe or worse non-proliferative, diabetic retinopathy in the study eye
4. Have history of vitrectomy, sub-macular surgery, or macular photocoagulation in the study eye
5. History of intraocular surgery in the study eye within 12 weeks prior to Visit 1
6. Have clinically significant cataract that may require surgery during the study period in the study eye
7. Presence of moderate to severe glaucomatous optic neuropathy, uncontrolled intraocular pressure (IOP), despite use of two or more topical agents; or a history of glaucoma-filtering or valve surgery
8. Axial myopia of greater than -8 diopters in the study eye
9. Have received any investigational product for the treatment of GA within the past 6 months or 5 half-lives (whichever is longer), other than nutritional supplements such as the age-related eye disease study (AREDS) formula
10. Have received a gene or cell therapy at any time.
11. Have a contraindication to the protocol specified corticosteroid regimen
12. Are unwilling to use two forms of contraception (one of which being a barrier method) for 90 days post-dosing, if relevant
13. Active malignancy within the past 12 months, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or prostate cancer with a stable prostate-specific antigen (PSA) ≥ 12 months
14. Have any other significant ocular or non-ocular medical or psychiatric condition which, in the opinion of the Investigator, may either put the subject at risk or may influence the results of the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (45):
  - Retinal Research Institute (retina consultants of AZ), Phoenix, Arizona
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Byers Eye Institute at Stanford, Palo Alto, California
  - Retina Consultants of San Diego, Poway, California
  - University of California (UC) Davis Medical Group Eye Center, Sacramento, California
  - Southwest Retina Research Center, Durango, Colorado
  - Rand Eye Institute, Deerfield Beach, Florida
  - VitreoRetinal Associates, P.A., Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Illinois Retina Associates, Chicago, Illinois
  - University Retina Macula Associates PC, Lemont, Illinois
  - Midwest Eye Institute Northside, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, LLC, Shawnee Mission, Kansas
  - The Retina Care Center, Baltimore, Maryland
  - Ophthalamic Consultants of Boston (OCB), Boston, Massachusetts
  - Retina Associates of Michigan, Grand Blanc, Michigan
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - Sierra Eye Associates, Reno, Nevada
  - Columbia University Medical Center, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - Duke Eye Center, Durham, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Retina, Eugene, Oregon
  - Casey Eye Institute - OHSU, Portland, Oregon
  - Erie Retinal Surgery ,INC, Erie, Pennsylvania
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Austin Research Center for Retina, PLLC, Austin, Texas
  - Retina Consultants of Houston-TMC, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Texas Retina Associates (Dallas), Dallas, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Department of Ophthalmology UW Medicine, Seattle, Washington
  - Retina Center Northwest, Silverdale, Washington
- Australia (2):
  - Sydney Hospital and Sydney Eye Hospital, Sydney, New South Wales
  - The University of Melbourne - The Centre for Eye Research Australia (CERA), Melbourne E., Victoria
- France (3):
  - CHU Dijon - Hopital Mitterrand, Dijon
  - Centre Paradis Monticelli, Marseille
  - CHU de Nantes - Hôtel-Dieu, Nantes
- Germany (4):
  - Universitätsklinikum Bonn, Bonn
  - Internationale Innovative Ophthalmochirurgie, Düsseldorf
  - Universitaetsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Universitaetsklinikum Tuebingen, Tübingen
- Oftalmika Spolka z ograniczona odpowiedzialnoscia, Bydgoszcz, Poland
- Spain (3):
  - Instituto de microcirugía ocular, Barcelona
  - Clinica Baviera, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
- United Kingdom (4):
  - Moorfields Eye Hospital - NHS Foundation Trust, London
  - Retina Clinic London, London
  - John Radcliffe Hospital, Oxford
  - Sunderland Eye Infirmary, Sunderland

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- See also: Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 3-arm study conducted in 2 stages. Results are reported per the 3 treatment arms. Stage 1 and Stage 2 results were combined since the study population and study treatments were the same in both Stage 1 and Stage 2; In Stage 1, participants were enrolled with both foveal and non-foveal geographic atrophy and in Stage 2, participants were enrolled with non-foveal geographic atrophy to enrich the number of participants with non-foveal geographic atrophy.
Pre-assignment Details: The study design with 3 arms was the same for both Stage 1 and 2. Analysis was performed following the statistical analysis plan to combine Stage 1 and 2 results, and to report results per the 3 unique treatment arms.
Period: Overall Study
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Started | 87 | 86 | 82
Stage 1 (Foveal and Non-foveal Geographic Atrophy) | 64 | 62 | 61
Stage 2 (Non-foveal Geographic Atrophy) | 23 | 24 | 21
Completed | 54 | 51 | 35
Not Completed | 33 | 35 | 47
Not completed — Death | 4 | 1 | 1
Not completed — Lost to Follow-up | 3 | 1 | 1
Not completed — Study terminated by sponsor | 11 | 17 | 32
Not completed — Withdrawal by Subject | 12 | 14 | 13
Not completed — Randomized but not treated due to AE | 2 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control | Total
Number analyzed (Participants) | 87 | 86 | 82 | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.6 (7.33) | 77.6 (7.60) | 77.8 (6.83) | 77.7 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 61 | 53 | 166
  Male | 35 | 25 | 29 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 87 | 80 | 80 | 247
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline to Week 72 in Geographic Atrophy (GA)
Description: GA area as measured by fundus autofluorescence (FAF)
Time Frame: Baseline, Weeks 12, 24, 36, 48 and 72
Population: Full Analysis Set - for participants with a valid measurement without a protocol deviation with impact.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 75 | 75 | 72
mm^2
  Week 12 (n=75,71,72): number analyzed (Participants) | 75 | 71 | 72
  Week 12 (n=75,71,72) | 0.730 (0.0625) | 0.752 (0.0634) | 0.667 (0.0647)
  Week 24 (n=72,75,71): number analyzed (Participants) | 72 | 75 | 71
  Week 24 (n=72,75,71) | 1.151 (0.0833) | 1.260 (0.0831) | 1.054 (0.0860)
  Week 36 (n=66,66,71): number analyzed (Participants) | 66 | 66 | 71
  Week 36 (n=66,66,71) | 1.728 (0.1488) | 1.955 (0.1503) | 1.531 (0.1528)
  Week 48 (n=64,68,65): number analyzed (Participants) | 64 | 68 | 65
  Week 48 (n=64,68,65) | 2.098 (0.1841) | 2.535 (0.1853) | 2.047 (0.1896)
  Week 72 (n=56,51,54): number analyzed (Participants) | 56 | 51 | 54
  Week 72 (n=56,51,54) | 3.225 (0.2337) | 3.421 (0.2369) | 2.919 (0.2412)
Statistical Analysis 1: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 12; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.062, 90% CI 2-sided [-0.087 to 0.211], Standard Error of Mean 0.0901
Statistical Analysis 2: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 12; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.084, 90% CI 2-sided [-0.066 to 0.234], Standard Error of Mean 0.0910
Statistical Analysis 3: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 24; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.096, 90% CI 2-sided [-0.102 to 0.294], Standard Error of Mean 0.1198
Statistical Analysis 4: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 24; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.205, 90% CI 2-sided [0.007 to 0.404], Standard Error of Mean 0.1200
Statistical Analysis 5: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 36; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.197, 90% CI 2-sided [-0.155 to 0.550], Standard Error of Mean 0.2135
Statistical Analysis 6: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 36; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.423, 90% CI 2-sided [0.068 to 0.779], Standard Error of Mean 0.2152
Statistical Analysis 7: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 48; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.052, 90% CI 2-sided [-0.385 to 0.489], Standard Error of Mean 0.2644
Statistical Analysis 8: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 48; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.488, 90% CI 2-sided [0.049 to 0.928], Standard Error of Mean 0.2662
Statistical Analysis 9: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 72; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.307, 90% CI 2-sided [-0.248 to 0.862], Standard Error of Mean 0.3361
Statistical Analysis 10: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 72; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.503, 90% CI 2-sided [-0.058 to 1.063], Standard Error of Mean 0.3392

2. Secondary Outcome: The Change From Baseline at Week 96 in Geographic Atrophy (GA)
Description: GA area as measured by fundus autofluorescence (FAF)
Time Frame: Baseline, Week 96
Population: Full Analysis Set - for participants with a valid measurement without a protocol deviation with impact.
Measure: Least Squares Mean (Standard Error); unit: mm2
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 44 | 39 | 32
mm2 | 4.414 (0.3109) | 4.607 (0.3167) | 3.769 (0.3286)
Statistical Analysis 1: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 96; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.645, 90% CI 2-sided [-0.103 to 1.393], Standard Error of Mean 0.4527
Statistical Analysis 2: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 96; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.838, 90% CI 2-sided [0.081 to 1.594], Standard Error of Mean 0.4577

3. Secondary Outcome: Summary of Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  A TEAE is defined as any AE that develops after randomization or any AE already present that worsens following randomization. The primary summaries of AEs are based on TEAEs.
Time Frame: Adverse events are reported from randomization to the end of study, at Week 96, up to a maximum timeframe of approximately 96 weeks.
Population: Full Analysis Set - all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 87 | 86 | 82
Participants
  Subjects with at least one ocular adverse event for the study eye | 66 | 65 | 15
  Subjects with at least one ocular adverse event for the fellow eye | 32 | 35 | 14
  Subjects with at least one non-ocular adverse event | 63 | 59 | 44
  Subjects with at least one ocular adverse event related to study treatment for the study eye | 13 | 21 | 0
  Subjects with at least one non-ocular adverse event related to study treatment | 0 | 0 | 0
  Subjects with at least one ocular adverse event related to surgical procedure for the study eye | 48 | 48 | 0
  Subjects with at least one non-ocular adverse event related to surgical procedure | 0 | 0 | 0
  Subjects with at least one ocular adverse event related to study procedure for the study eye | 8 | 9 | 0
  Subjects with at least one non-ocular adverse event related to study procedure | 0 | 2 | 0
  Subjects with at least one ocular adverse event leading to study discontinuation for the study eye | 0 | 0 | 0
  Subjects with at least one non-ocular adverse event leading to study discontinuation | 5 | 2 | 1
  Subjects with at least one ocular adverse event of special interest for the study eye | 19 | 31 | 3
  Subjects with at least one ocular adverse event of special interest for the fellow eye | 3 | 3 | 1
  Subjects with at least one ocular serious adverse event (SAE) for the study eye | 2 | 5 | 0
  Subjects with at least one ocular serious adverse event for the fellow eye | 0 | 0 | 0
  Subjects with at least one non-ocular serious adverse event | 20 | 22 | 10
  Subjects with at least one ocular serious adverse event related to study treatment for the study eye | 0 | 0 | 0
  Subjects with at least one non-ocular serious adverse event related to study treatment | 0 | 0 | 0
  Subjects with at least one ocular SAE related to surgical procedure for the study eye | 1 | 4 | 0
  Subjects with at least one non-ocular serious adverse event related to surgical procedure | 0 | 0 | 0
  Subjects with at least one ocular serious adverse event related to study procedure for the study eye | 1 | 1 | 0
  Subjects with at least one non-ocular serious adverse event related to study procedure | 0 | 0 | 0
  Subjects with at least one ocular SAE leading to study discontinuation for the study eye | 0 | 0 | 0
  Subjects with at least one non-ocular serious adverse event leading to study discontinuation | 5 | 2 | 1
  Deaths | 4 | 1 | 1

4. Secondary Outcome: Ocular AEs Occurring in ≥2% of Subjects by Primary System Organ Class and Preferred Term for the Study Eye
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  A TEAE is defined as any AE that develops after randomization or any AE already present that worsens following randomization. The primary summaries of AEs are based on TEAEs.
  System organ classes are sorted alphabetically, and preferred terms are sorted by decreasing overall frequency within system organ class.
Time Frame: as for outcome 3
Population: Full Analysis Set - all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 87 | 86 | 82
Participants
  Subjects with at least one event | 66 | 65 | 15
  Eye disorders | 65 | 62 | 14
  -Cataract | 21 | 20 | 3
  -Retinal pigmentation | 12 | 22 | 0
  -Conjunctival haemorrhage | 18 | 12 | 1
  -Retinal haemorrhage | 8 | 10 | 2
  -Eye pain | 5 | 7 | 0
  -Ocular hypertension | 6 | 6 | 0
  -Punctate keratitis | 6 | 6 | 0
  -Retinal tear | 5 | 6 | 0
  -Dry eye | 4 | 4 | 1
  -Posterior capsule opacification | 3 | 4 | 2
  -Anterior chamber cell | 4 | 4 | 0
  -Eye irritation | 6 | 2 | 0
  -Vitreous haemorrhage | 2 | 6 | 0
  -Choroidal neovascularisation | 2 | 3 | 2
  -Vitreous floaters | 3 | 4 | 0
  -Cataract nuclear | 3 | 3 | 0
  -Retinal detachment | 2 | 4 | 0
  -Corneal oedema | 1 | 4 | 0
  -Diplopia | 4 | 1 | 0
  -Eye pruritus | 1 | 4 | 0
  -Foreign body sensation in eyes | 3 | 2 | 0
  -Iritis | 4 | 1 | 0
  -Visual impairment | 2 | 3 | 0
  Investigations | 11 | 2 | 0
  -Intraocular pressure increased | 1 | 2 | 0

5. Secondary Outcome: Non-ocular AEs Occurring in ≥2% of Subjects
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Full Analysis Set - all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 87 | 86 | 82
Participants | 63 | 59 | 44

6. Secondary Outcome: Change in GA Morphology From Baseline to Week 96 on Multimodal Imaging - Number of Participants With Increase in Fundus Autofluorescence
Description: Change in retinal morphology on multimodal imaging.
  For the untreated control group, there were no protocol-specified visits at Week 5.
Time Frame: Baseline, Weeks 5, 12, 24, 36, 48, 72 and 96
Population: Full Analysis Set - for participants with a valid measurement without a protocol deviation with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 75 | 78 | 74
Participants
  Week 5 (n=23,24,0): number analyzed (Participants) | 23 | 24 | 0
  Week 5 (n=23,24,0) | 23 | 23 |
  Week 12 (n=75,73,74): number analyzed (Participants) | 75 | 73 | 74
  Week 12 (n=75,73,74) | 74 | 73 | 73
  Week 24 (n=75,78,72): number analyzed (Participants) | 75 | 78 | 72
  Week 24 (n=75,78,72) | 72 | 78 | 71
  Week 36 (n=70,70, 71): number analyzed (Participants) | 70 | 70 | 71
  Week 36 (n=70,70, 71) | 66 | 69 | 70
  Week 48 (n=67,72,68): number analyzed (Participants) | 67 | 72 | 68
  Week 48 (n=67,72,68) | 67 | 71 | 68
  Week 72 (n=61, 62,59): number analyzed (Participants) | 61 | 62 | 59
  Week 72 (n=61, 62,59) | 60 | 60 | 56
  Week 96 (n=52,49, 34): number analyzed (Participants) | 52 | 49 | 34
  Week 96 (n=52,49, 34) | 50 | 48 | 33

7. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) Score From Baseline Through Week 96 Via the Early Treatment for Diabetic Retinopathy (ETDRS) Chart
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
  For the untreated control group, there were no protocol-specified visits for Weeks 1, 5 and 8.
Time Frame: Baseline, Weeks 1, 5, 8, 12, 24, 36, 48, 72 and 96
Population: Full Analysis Set - for participants with a valid measurement without a protocol deviation with impact.
Measure: Least Squares Mean (Standard Error); unit: Letters read
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 81 | 79 | 73
Letters read
  Week 1 (n=81,78,0): number analyzed (Participants) | 81 | 78 | 0
  Week 1 (n=81,78,0) | -2.0 (1.54) | -7.0 (1.56) |
  Week 5 (n=81,78,0): number analyzed (Participants) | 81 | 78 | 0
  Week 5 (n=81,78,0) | -0.8 (0.88) | -3.3 (0.89) |
  Week 8 (n=79,77,0): number analyzed (Participants) | 79 | 77 | 0
  Week 8 (n=79,77,0) | -0.1 (0.85) | -1.7 (0.86) |
  Week 12 (n=79,79,73): number analyzed (Participants) | 79 | 79 | 73
  Week 12 (n=79,79,73) | -1.1 (0.91) | -2.5 (0.91) | -0.7 (0.96)
  Week 24 (n=78,78,71): number analyzed (Participants) | 78 | 78 | 71
  Week 24 (n=78,78,71) | -2.7 (1.03) | -6.3 (1.03) | -1.1 (1.09)
  Week 36 (75,74,72): number analyzed (Participants) | 75 | 74 | 72
  Week 36 (75,74,72) | -2.5 (1.24) | -7.7 (1.25) | -3.0 (1.30)
  Week 48 (n=73,75,69): number analyzed (Participants) | 73 | 75 | 69
  Week 48 (n=73,75,69) | -2.6 (1.48) | -7.3 (1.46) | -5.3 (1.54)
  Week 72 (n=63, 70, 58): number analyzed (Participants) | 63 | 70 | 58
  Week 72 (n=63, 70, 58) | -4.1 (1.54) | -7.9 (1.50) | -8.8 (1.61)
  Week 96 (n=54,51,35): number analyzed (Participants) | 54 | 51 | 35
  Week 96 (n=54,51,35) | -5.5 (1.78) | -10.0 (1.78) | -12.7 (2.02)
Statistical Analysis 1: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 12; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -0.5, 90% CI 2-sided [-2.6 to 1.7], Standard Error of Mean 1.33
Statistical Analysis 2: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 12; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -1.8, 90% CI 2-sided [-4.0 to 0.4], Standard Error of Mean 1.32
Statistical Analysis 3: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 24; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -1.6, 90% CI 2-sided [-4.1 to 0.8], Standard Error of Mean 1.50
Statistical Analysis 4: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 24; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -5.3, 90% CI 2-sided [-7.7 to -2.8], Standard Error of Mean 1.49
Statistical Analysis 5: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 36; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.5, 90% CI 2-sided [-2.5 to 3.5], Standard Error of Mean 1.81
Statistical Analysis 6: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 36; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -4.7, 90% CI 2-sided [-7.7 to -1.7], Standard Error of Mean 1.80
Statistical Analysis 7: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 48; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 2.6, 90% CI 2-sided [-0.9 to 6.1], Standard Error of Mean 2.14
Statistical Analysis 8: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 48; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -2.1, 90% CI 2-sided [-5.6 to 1.4], Standard Error of Mean 2.12
Statistical Analysis 9: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 72; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 4.7, 90% CI 2-sided [1.0 to 8.4], Standard Error of Mean 2.24
Statistical Analysis 10: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 72; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.9, 90% CI 2-sided [-2.8 to 4.5], Standard Error of Mean 2.20
Statistical Analysis 11: Comparison: GT005 Medium Dose [5E10 vg] vs Untreated Control; Week 96; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 7.1, 90% CI 2-sided [2.7 to 11.6], Standard Error of Mean 2.70
Statistical Analysis 12: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 96; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 2.6, 90% CI 2-sided [-1.8 to 7.1], Standard Error of Mean 2.68

8. Secondary Outcome: Change in Low Luminance Difference (LLD) Letter Count From Baseline at Weeks 12, 24, 36, 48, 72 and 96, Via Early Treatment for Diabetic Retinopathy (ETDRS) Chart
Description: LLD was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  The test was to be performed after BCVA testing, prior to pupil dilation, and distance refraction was to be carried out before Low Luminance Visual Acuity (LLVA) was measured.
  LLVA was to be measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the subject read the normally illuminated ETDRS chart. The LLD was calculated as the difference between BCVA and LLVA.
  Initially, letters were to be read at a distance of 4 metres from the chart. If <20 letters were read at 4 metres, testing at 1 metre should have been performed. LLD was to be reported as number of letters read correctly by the subject.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72 and 96
Population: Full Analysis Set - for participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 79 | 76 | 74
Letters read
  Week 12 | -0.6 (7.59) | -1.1 (9.63) | 1.2 (9.51)
  Week 24 (n=78,75,71): number analyzed (Participants) | 78 | 75 | 71
  Week 24 (n=78,75,71) | -0.6 (10.10) | -2.5 (12.73) | 0.5 (12.01)
  Week 36 (n=75,72,71): number analyzed (Participants) | 75 | 72 | 71
  Week 36 (n=75,72,71) | 0.0 (9.90) | -2.6 (13.40) | -0.1 (11.12)
  Week 48 (n=73,73,69): number analyzed (Participants) | 73 | 73 | 69
  Week 48 (n=73,73,69) | -0.5 (10.31) | -1.5 (15.18) | -0.4 (12.93)
  Week 72 (n=63,67,58): number analyzed (Participants) | 63 | 67 | 58
  Week 72 (n=63,67,58) | -0.5 (13.15) | -5.2 (17.24) | -2.5 (14.93)
  Week 96 (n=54,49,35): number analyzed (Participants) | 54 | 49 | 35
  Week 96 (n=54,49,35) | -3.1 (16.11) | -2.2 (13.48) | -5.9 (16.82)

9. Secondary Outcome: Reading Performance, Measured as the MRS (Words Per Minute), as Assessed by Minnesota Low-vision Reading Test (MNRead) Chart: Summary Statistics for Change From Baseline by Visit for the Study Eye
Description: The maximum reading speed (MRS) represents the highest reading speed an individual can achieve when print size is not a limiting factor. Essentially, it measures how quickly a person can read text when the print is large enough to be easily readable.
  A higher count represents better visual functioning.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72 and 96
Population: Full Analysis Set - for participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Words read per minute
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 73 | 72 | 65
Words read per minute
  Week 24 (n=73,72,65) | -15.756 (32.7268) | -12.368 (43.2054) | -15.769 (40.5051)
  Week 36 (n=71,70,65): number analyzed (Participants) | 71 | 70 | 65
  Week 36 (n=71,70,65) | -18.488 (54.7913) | -15.673 (31.7802) | -3.689 (94.1057)
  Week 48 (n=69,67,62): number analyzed (Participants) | 69 | 67 | 62
  Week 48 (n=69,67,62) | -20.734 (36.4110) | -6.678 (49.0844) | -17.297 (56.8547)
  Week 72 (n=57,64,53): number analyzed (Participants) | 57 | 64 | 53
  Week 72 (n=57,64,53) | -24.485 (45.8525) | -20.798 (39.6796) | -26.121 (40.8016)
  Week 96 (n=48,47,29): number analyzed (Participants) | 48 | 47 | 29
  Week 96 (n=48,47,29) | -24.678 (44.7777) | -25.178 (39.7216) | -19.242 (45.0703)

10. Secondary Outcome: Change From Baseline at Weeks 24, 36, 48, 72 and 96 in Functional Reading Independence (FRI) Index
Description: The FRI index is a patient-reported outcome measure developed specifically for use in GA patients. The FRI index evaluates the level of independence subjects have in performing everyday activities that require reading, such as writing a cheque or reading a prescription.
  Scores derived from the index range from 1 (unable to do) to 4 (total independence).
  A higher score represents better visual functioning.
Time Frame: Baseline, Weeks 24, 36, 48, 72 and 96
Population: Full Analysis Set - for participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 77 | 75 | 67
Scores on a scale
  Week 24 (n=77,75,67) | -0.4 (5.20) | -1.4 (4.74) | -0.1 (3.98)
  Week 36 (n=74,72,66): number analyzed (Participants) | 74 | 72 | 66
  Week 36 (n=74,72,66) | -0.8 (4.64) | -1.1 (4.31) | -0.1 (4.67)
  Week 48 (n=70,73,65): number analyzed (Participants) | 70 | 73 | 65
  Week 48 (n=70,73,65) | -0.3 (4.76) | -1.4 (4.87) | -0.2 (4.50)
  Week 72 (n=63,69,58): number analyzed (Participants) | 63 | 69 | 58
  Week 72 (n=63,69,58) | -0.8 (4.93) | -1.3 (5.19) | -1.5 (5.37)
  Week 96 (n=54,51,32): number analyzed (Participants) | 54 | 51 | 32
  Week 96 (n=54,51,32) | -1.4 (5.57) | -1.4 (4.41) | -1.1 (5.11)

11. Secondary Outcome: Change From Baseline at Weeks 24, 36, 48, 72 and 96 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Composite Score
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) measures the influence of visual disability and visual symptoms on general health domains.
  The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better visual functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. A composite score is derived based on the average of the 11 subscales.
Time Frame: Baseline, Weeks 24, 36, 48, 72 and 96
Population: Full Analysis Set - for participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GT005 Medium Dose [5E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 77 | 78 | 67
Scores on a scale
  Week 24 (n=77,78,67) | -1.466 (12.8742) | -2.289 (12.3295) | -1.270 (11.2063)
  Week 36 (n=74,73,66): number analyzed (Participants) | 74 | 73 | 66
  Week 36 (n=74,73,66) | -1.955 (11.5060) | -3.479 (12.0848) | -2.273 (12.2395)
  Week 48 (n=70,74,65): number analyzed (Participants) | 70 | 74 | 65
  Week 48 (n=70,74,65) | -2.501 (12.9563) | -3.113 (11.9974) | -4.403 (14.2465)
  Week 72 (n=63,69,54): number analyzed (Participants) | 63 | 69 | 54
  Week 72 (n=63,69,54) | -4.232 (14.6259) | -3.432 (11.3840) | -6.583 (15.5133)
  Week 96 (n=54,51,33): number analyzed (Participants) | 54 | 51 | 33
  Week 96 (n=54,51,33) | -6.341 (14.4187) | -7.718 (10.9016) | -6.804 (15.4812)

ADVERSE EVENTS:
Time Frame: Adverse events are reported from randomization to the end of study, at Week 96, up to a maximum timeframe of approximately 96 weeks.
Groups:
- GT005@Medium Dose@[5E10 vg]: GT005@Medium dose@[5E10 vg]
- GT005@High Dose@[2E11 vg]: GT005@High dose@[2E11 vg]
- Overall: Overall
Arm/Group | GT005@Medium Dose@[5E10 vg] | GT005@High Dose@[2E11 vg] | Untreated Control | Overall
All-Cause Mortality (participants affected / at risk) | 4/87 | 1/86 | 1/82 | 6/255
Serious Adverse Events (participants affected / at risk) | 22/87 | 25/86 | 10/82 | 57/255
Other Adverse Events (participants affected / at risk) | 76/87 | 75/86 | 50/82 | 201/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GT005@Medium Dose@[5E10 vg] (N=87) | GT005@High Dose@[2E11 vg] (N=86) | Untreated Control (N=82) | Overall (N=255)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 0 | 4
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 0 | 2
Chronic left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 1
Coronary artery dissection (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 1 | 3
Retinal detachment - Study eye (Eye disorders) | 1 | 2 | 0 | 3
Vitreous haemorrhage - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 1 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 2
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1
Endophthalmitis - Study eye (Infections and infestations) | 0 | 3 | 0 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2
Pneumonia serratia (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 2 | 0 | 3
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Dural tear (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Open globe injury - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Sarcomatoid carcinoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 1 | 3
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Embolic stroke (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 1 | 0 | 3
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GT005@Medium Dose@[5E10 vg] (N=87) | GT005@High Dose@[2E11 vg] (N=86) | Untreated Control (N=82) | Overall (N=255)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 8
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Aortic valve calcification (Cardiac disorders) | 1 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 1 | 6
Cardiac amyloidosis (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 2
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 2
Left ventricular failure (Cardiac disorders) | 0 | 2 | 1 | 3
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Corneal dystrophy - Fellow eye (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1
Corneal dystrophy - Study eye (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 2
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 3
Anterior capsule contraction - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Anterior capsule contraction - Study eye (Eye disorders) | 0 | 0 | 1 | 1
Anterior chamber cell - Study eye (Eye disorders) | 4 | 4 | 0 | 8
Anterior chamber flare - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Blepharitis - Fellow eye (Eye disorders) | 2 | 0 | 0 | 2
Blepharitis - Study eye (Eye disorders) | 3 | 1 | 0 | 4
Borderline glaucoma - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Borderline glaucoma - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Cataract - Fellow eye (Eye disorders) | 5 | 10 | 2 | 17
Cataract - Study eye (Eye disorders) | 21 | 20 | 3 | 44
Cataract nuclear - Fellow eye (Eye disorders) | 2 | 0 | 0 | 2
Cataract nuclear - Study eye (Eye disorders) | 3 | 3 | 0 | 6
Cataract subcapsular - Fellow eye (Eye disorders) | 0 | 1 | 0 | 1
Cataract subcapsular - Study eye (Eye disorders) | 1 | 2 | 0 | 3
Chalazion - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Chalazion - Study eye (Eye disorders) | 3 | 1 | 0 | 4
Choroidal detachment - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Choroidal haemorrhage - Study eye (Eye disorders) | 1 | 1 | 0 | 2
Choroidal neovascularisation - Fellow eye (Eye disorders) | 1 | 1 | 1 | 3
Choroidal neovascularisation - Study eye (Eye disorders) | 2 | 3 | 2 | 7
Chromatopsia - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Conjunctival haemorrhage - Study eye (Eye disorders) | 18 | 12 | 1 | 31
Conjunctival oedema - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Corneal defect - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Corneal disorder - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Corneal epithelial microcysts - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Corneal erosion - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Corneal oedema - Fellow eye (Eye disorders) | 0 | 1 | 0 | 1
Corneal oedema - Study eye (Eye disorders) | 1 | 4 | 0 | 5
Corneal striae - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Cystoid macular oedema - Study eye (Eye disorders) | 1 | 2 | 0 | 3
Dermatochalasis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Detachment of retinal pigment epithelium - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Diplopia - Fellow eye (Eye disorders) | 3 | 1 | 0 | 4
Diplopia - Study eye (Eye disorders) | 4 | 1 | 0 | 5
Dry age-related macular degeneration - Fellow eye (Eye disorders) | 2 | 0 | 0 | 2
Dry eye - Fellow eye (Eye disorders) | 2 | 4 | 1 | 7
Dry eye - Study eye (Eye disorders) | 4 | 4 | 1 | 9
Ectropion - Fellow eye (Eye disorders) | 0 | 2 | 1 | 3
Ectropion - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Eczema eyelids - Fellow eye (Eye disorders) | 2 | 0 | 0 | 2
Eczema eyelids - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Epiretinal membrane - Study eye (Eye disorders) | 1 | 1 | 0 | 2
Exophthalmos - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Eye discharge - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Eye inflammation - Study eye (Eye disorders) | 0 | 2 | 0 | 2
Eye irritation - Study eye (Eye disorders) | 6 | 2 | 0 | 8
Eye pain - Study eye (Eye disorders) | 5 | 7 | 0 | 12
Eye pruritus - Study eye (Eye disorders) | 1 | 4 | 0 | 5
Eyelid bleeding - Study eye (Eye disorders) | 2 | 1 | 0 | 3
Eyelid oedema - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Eyelid pain - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Eyelid ptosis - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Eyelids pruritus - Fellow eye (Eye disorders) | 1 | 1 | 0 | 2
Eyelids pruritus - Study eye (Eye disorders) | 2 | 1 | 0 | 3
Foreign body sensation in eyes - Study eye (Eye disorders) | 3 | 2 | 0 | 5
Foveal degeneration - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Fuchs' syndrome - Fellow eye (Eye disorders) | 0 | 1 | 0 | 1
Fuchs' syndrome - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Glare - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Glaucoma - Fellow eye (Eye disorders) | 1 | 2 | 0 | 3
Glaucoma - Study eye (Eye disorders) | 2 | 2 | 0 | 4
Hypotony of eye - Study eye (Eye disorders) | 1 | 1 | 0 | 2
Iridocyclitis - Study eye (Eye disorders) | 1 | 3 | 0 | 4
Iritis - Study eye (Eye disorders) | 4 | 1 | 0 | 5
Keratic precipitates - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Keratitis - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Keratitis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Lacrimation decreased - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Lacrimation decreased - Study eye (Eye disorders) | 0 | 0 | 1 | 1
Lacrimation disorder - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Lacrimation increased - Study eye (Eye disorders) | 1 | 1 | 0 | 2
Lagophthalmos - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Lens dislocation - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Lenticular opacities - Study eye (Eye disorders) | 0 | 1 | 1 | 2
Macular hole - Study eye (Eye disorders) | 0 | 0 | 1 | 1
Macular oedema - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Metamorphopsia - Fellow eye (Eye disorders) | 0 | 1 | 0 | 1
Metamorphopsia - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 2 | 2 | 1 | 5
Ocular discomfort - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Ocular discomfort - Study eye (Eye disorders) | 2 | 2 | 0 | 4
Ocular hyperaemia - Study eye (Eye disorders) | 1 | 1 | 0 | 2
Ocular hypertension - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Ocular hypertension - Study eye (Eye disorders) | 6 | 6 | 0 | 12
Optic disc haemorrhage - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Optic ischaemic neuropathy - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Optic ischaemic neuropathy - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Optic nerve sheath haemorrhage - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Periorbital pain - Study eye (Eye disorders) | 2 | 0 | 0 | 2
Photophobia - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Photopsia - Fellow eye (Eye disorders) | 0 | 1 | 0 | 1
Photopsia - Study eye (Eye disorders) | 2 | 2 | 0 | 4
Posterior capsule opacification - Fellow eye (Eye disorders) | 5 | 4 | 2 | 11
Posterior capsule opacification - Study eye (Eye disorders) | 3 | 4 | 2 | 9
Pterygium - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Punctate keratitis - Fellow eye (Eye disorders) | 4 | 6 | 0 | 10
Punctate keratitis - Study eye (Eye disorders) | 6 | 6 | 0 | 12
Retinal cyst - Fellow eye (Eye disorders) | 0 | 1 | 0 | 1
Retinal depigmentation - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Retinal depigmentation - Study eye (Eye disorders) | 1 | 1 | 0 | 2
Retinal detachment - Study eye (Eye disorders) | 1 | 2 | 0 | 3
Retinal haemorrhage - Fellow eye (Eye disorders) | 1 | 2 | 0 | 3
Retinal haemorrhage - Study eye (Eye disorders) | 8 | 10 | 2 | 20
Retinal oedema - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Retinal pigmentation - Fellow eye (Eye disorders) | 1 | 1 | 0 | 2
Retinal pigmentation - Study eye (Eye disorders) | 12 | 22 | 0 | 34
Retinal tear - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Retinal tear - Study eye (Eye disorders) | 5 | 6 | 0 | 11
Retinal vein occlusion - Study eye (Eye disorders) | 1 | 0 | 1 | 2
Subretinal fluid - Study eye (Eye disorders) | 2 | 0 | 0 | 2
Swelling of eyelid - Study eye (Eye disorders) | 2 | 0 | 0 | 2
Tractional retinal detachment - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Trichiasis - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Trichiasis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Ulcerative keratitis - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Vision blurred - Study eye (Eye disorders) | 2 | 0 | 0 | 2
Visual field defect - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Visual impairment - Fellow eye (Eye disorders) | 1 | 2 | 0 | 3
Visual impairment - Study eye (Eye disorders) | 2 | 3 | 0 | 5
Vitreal cells - Study eye (Eye disorders) | 2 | 0 | 0 | 2
Vitreoretinal traction syndrome - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Vitreous detachment - Fellow eye (Eye disorders) | 1 | 1 | 2 | 4
Vitreous floaters - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Vitreous floaters - Study eye (Eye disorders) | 3 | 4 | 0 | 7
Vitreous haemorrhage - Fellow eye (Eye disorders) | 0 | 1 | 0 | 1
Vitreous haemorrhage - Study eye (Eye disorders) | 2 | 6 | 0 | 8
Vitreous opacities - Study eye (Eye disorders) | 2 | 1 | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 4 | 0 | 5
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 3 | 0 | 6
Oesophageal dysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 3 | 0 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Chest pain (General disorders) | 1 | 0 | 0 | 1
Discomfort (General disorders) | 1 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 0 | 1
Facial pain - Study eye (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 1 | 4
Illness (General disorders) | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 1 | 2
Infusion site bruising (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 2
Prosthetic cardiac valve stenosis (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 2
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 2 | 0 | 2
Abscess intestinal (Infections and infestations) | 0 | 1 | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1 | 2 | 5
COVID-19 (Infections and infestations) | 14 | 12 | 9 | 35
Candida infection (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2 | 0 | 4
Conjunctivitis - Fellow eye (Infections and infestations) | 2 | 0 | 0 | 2
Conjunctivitis - Study eye (Infections and infestations) | 2 | 1 | 0 | 3
Conjunctivitis bacterial - Fellow eye (Infections and infestations) | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 3 | 0 | 0 | 3
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 2
Eye infection - Fellow eye (Infections and infestations) | 0 | 0 | 1 | 1
Eye infection - Study eye (Infections and infestations) | 0 | 0 | 1 | 1
Eyelid infection - Fellow eye (Infections and infestations) | 0 | 1 | 0 | 1
Furuncle (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 1
Gingival abscess (Infections and infestations) | 0 | 0 | 1 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1
Hordeolum - Fellow eye (Infections and infestations) | 0 | 1 | 0 | 1
Hordeolum - Study eye (Infections and infestations) | 1 | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 2 | 0 | 2
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 1
Leprosy (Infections and infestations) | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Lyme disease (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 4 | 0 | 5
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 1 | 5 | 0 | 6
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Pyuria (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1
Root canal infection (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 4 | 1 | 6
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 3 | 1 | 4
Tooth infection (Infections and infestations) | 2 | 1 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 3
Urinary tract infection (Infections and infestations) | 7 | 3 | 3 | 13
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Accidental exposure to product - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Chemical burns of eye - Fellow eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Chemical burns of eye - Study eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Corneal abrasion - Study eye (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Craniofacial fracture - Fellow eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Eye contusion - Study eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Eyelid contusion - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Eyelid injury - Fellow eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 5
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Hyphaema - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural pain - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Product administered at inappropriate site - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Retinal tear - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Skin laceration - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Splinter (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Suture related complication - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 2 | 4
Blood creatinine increased (Investigations) | 3 | 0 | 0 | 3
Blood glucose increased (Investigations) | 1 | 1 | 0 | 2
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 1
Blood pressure increased (Investigations) | 3 | 0 | 3 | 6
Blood pressure systolic increased (Investigations) | 1 | 0 | 1 | 2
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 5 | 2 | 2 | 9
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 1
Full blood count abnormal (Investigations) | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 1 | 0 | 2
Haemoglobin decreased (Investigations) | 0 | 2 | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 1
Intraocular pressure increased - Fellow eye (Investigations) | 1 | 1 | 0 | 2
Intraocular pressure increased - Study eye (Investigations) | 11 | 2 | 0 | 13
Lipase increased (Investigations) | 2 | 4 | 0 | 6
Liver function test increased (Investigations) | 1 | 0 | 0 | 1
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 1 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1 | 1 | 2
Platelet count decreased (Investigations) | 2 | 0 | 0 | 2
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 0 | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 1 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 7
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 5
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1 | 5
Basal cell carcinoma - Study eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Eye naevus - Study eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Amputation stump pain (Nervous system disorders) | 0 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral atrophy (Nervous system disorders) | 1 | 0 | 1 | 2
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 1 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 1 | 1 | 2
Gerstmann's syndrome (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 5 | 0 | 6
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Ilioinguinal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 1 | 1
Neuralgia - Fellow eye (Nervous system disorders) | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 2 | 0 | 2
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 1 | 1 | 2
VIth nerve paralysis - Study eye (Nervous system disorders) | 0 | 1 | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 1
Device dislocation - Study eye (Product Issues) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 3
Charles Bonnet syndrome (Psychiatric disorders) | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 2
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 1
Glomerulosclerosis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1
Microalbuminuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 2 | 5
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 2 | 3
Ureteric dilatation (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin mass - Study eye (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Edentulous (Social circumstances) | 1 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 4 | 4 | 1 | 9
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 1 | 3
Lymphocele (Vascular disorders) | 0 | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
White coat hypertension (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04566445/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT04566445/SAP_001.pdf